CLINICAL TRIAL: NCT06083337
Title: Vascular Inflammation ReDuction and Perivascular Fat Imaging by Computed Tomography
Acronym: VIRDICT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hippocration General Hospital (Other)
Collaborators: Biomedical Research Foundation, Academy of Athens (Other)
Responsible Party: Principal Investigator, Alexios S. Antonopoulos, Academic Consultant Cardiologist, Non-Invasive Imaging Specialist (CT/CMR), Hippocration General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 7121/29-11-2018/00468
Record Dates: First submitted 2023-10-05; First posted 2023-10-16 (Actual); Last update posted 2023-10-16 (Actual); Status verified 2023-10

CONDITIONS: Coronary Artery Disease; Atheroscleroses, Coronary; Vascular Inflammation
Keywords: vascular inflammation; fat attenuation index; pericoronary adipose tissue; coronary computed tomography angiography
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Intervention Model Description: Participants of the VIRDICT study will be randomized either to standard of care management or high-dose atorvastatin +/- colchicine.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard of care management (No Intervention): Patients will receive standard of care treatment.
- Coronary inflammation-based management (Experimental): Participants classified as moderate risk (FAI-Score 75th-89th percentile for the RCA or the LAD or ≥ 95th percentile for the LCx) or CaRi-Heart risk≥ 5% and <10%) will receive atorvastatin 40mg daily, if they do not already receive statin therapy, while if they already receive statin, it will be discontinued and they will be given atorvastatin 80 mg daily. Participants classified as high risk (FAI-Score≥ 90th percentile for the RCA or the LAD or CaRi-Heart risk≥ 10%) will receive atorvastatin 80 mg daily and colchicine 0.5 mg daily. Tolerance and compliance will be monitored during the study follow-up and participants will be informed at enrollment about possible treatment side effects. In case of colchicine intolerance, colchicine will be discontinued. If the patient cannot tolerate atorvastatin, then half dose may be prescribed daily. In case of severe adverse events related to atorvastatin, atorvastatin will be discontinued and the participant will withdraw from the study.
  Interventions: Device: CaRi-Heart device

INTERVENTIONS:
Device: CaRi-Heart device — Open-label treatment with atorvastatin +/- low-dose colchicine medications based on CaRi-Heart algorithm management.
  Arms: Coronary inflammation-based management

SUMMARY:
The goal of this clinical trial is to compare the effect of standard of care management vs. CaRi-Heart based management on vascular inflammation in patients with increased Fat Attenuation Index-Score. The main questions it aims to answer are:

* Does treatment intensification reduce vascular inflammation detected by perivascular fat imaging to a greater extent than standard of care treatment?
* Do changes in vascular inflammation biomarkers correlate with changes in lipid metrics or inflammatory biomarkers, such as interleukin-6?

Participants will be randomized either to standard of care treatment or intensified treatment with maximum dose of atorvastatin +/- low dose of colchicine. After their inclusion, study participants will be followed-up for 6 months with regular monitoring for adverse events and blood will be drawn at 3 and 6 months. After the 6-month follow-up, participants will undergo CCTA imaging for fat attenuation index measurements. Researchers will compare standard of care and vascular inflammation-based treatment to see if inflammation-based treatment is more potent against vascular inflammation.

DETAILED DESCRIPTION:
The VIRDICT study is a randomized, open-label clinical study including participants aged 30-80 years old, who underwent coronary computed tomography angiography (CCTA) and had no obstructive coronary stenoses. CCTA images will be transferred as pseudonymized DICOM data to Caristo Diagnostics Ltd for perivascular fat analysis. Individuals with evidence of coronary inflammation, as assessed by fat attenuation index (FAI) will be eligible for the VIRDICT study. Participants will be randomized either to standard of care treatment or inflammation-based treatment with atorvastatin ± colchicine. Participants will be followed-up for 6 months post randomization, with four follow-up visits (two by telephone call and two by onsite visit). At the end of their follow-up, participants will undergo a second CCTA and the relevant images will be analyzed for pericoronary inflammation. 140 participants are expected be included in the study. Interim analyses will be performed after sufficient patients (approximately 80 patients) have completed 24 weeks of follow-up. This is a pilot study to establish the ability of CCTA-derived FAI quantification to detect a change in coronary artery inflammation, following a period of treatment with medications with known anti-inflammatory properties (statin and colchicine).

ELIGIBILITY:
Inclusion Criteria:

Participants must satisfy the following conditions:

1. Male or female, aged 30 to 80 years
2. CCTA scan showing mild coronary artery plaques (<50% luminal stenosis) and CaRi-Heart Risk ≥ 5% and/or FAI-Score ≥ 75th percentile in the left anterior coronary or right coronary artery or FAI-Score ≥ 95th percentile in the circumflex coronary within the last 6 months.
3. Willing and able (in the Investigators opinion) to comply with all study requirements.
4. Able to understand both verbal or written Greek
5. No definite clinical indication for a change in treatment based on European Society of Cardiology guidelines or planned revascularization

Exclusion Criteria:

The participant may not enter the study if ANY of the following are known to apply:

1. Previous documented history of coronary artery disease requiring treatment. This includes any of the following:

   i. Acute myocardial infarction ii. Unstable angina iii. Coronary revascularization procedure iv. Clinically significant coronary artery disease diagnosed by invasive or non-invasive testing.
2. History of New York Heart Association (NYHA) Class III or IV heart failure within the past 12 months of consent.
3. Autoimmune disease requiring immunosuppressive therapy or systemic corticosteroid therapy
4. Active chronic treatment with any anti-inflammatory agents (e.g. NSAIDs, systemic corticosteroids)
5. Active neoplasm requiring surgery, chemotherapy, or radiation within the prior 12 months (subjects with a history of malignancy who have undergone curative resection or otherwise not requiring treatment for at least 12 months prior to screening with no detectable recurrence are allowed)
6. Contraindication for statin therapy. Patients with intolerance to colchicine therapy may be included but they will receive statin treatment only.
7. Severe Chronic kidney disease (estimated glomerular filtration rate < 30 mL/min/1.73 m² and/or serum creatinine > 2.5 mg/dL or 220 µmol/l).
8. Hepatic dysfunction (aspartate aminotransferase [AST] or alanine aminotransferase [ALT] > 3 × the upper limit of normal [ULN] measured on local labs in last 6 months)
9. Any clinically significant abnormality identified at the time of screening that, in the opinion of the Investigator, would preclude safe completion of the study.
10. Any other significant disease or disorder which, in the opinion of the Investigator, may either put the participants at risk because of participation in the study, or may influence the result of the study, or the participant's ability to participate in the study.
11. Participants who have participated in another research study involving a treatment intervention or an investigational product, in the past 12 weeks.
12. Patients unable to understand verbal or written English.
13. Contraindication to contract dye for CCTA.
14. Pregnancy

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2022-01-22 (Actual); Primary Completion 2025-07-22 (Estimated); Study Completion 2025-07-22 (Estimated)

PRIMARY OUTCOMES:
Change in Fat Attenuation Index (FAI) in the proximal right coronary (RCA), left anterior descending (LAD) and circumflex (Cx) coronary arteries | 6 months
  FAI change will be compared between the standard of care arm and the inflammation-based treatment arm

SECONDARY OUTCOMES:
% change in plasma LDL-c | 6 months
  Change in LDL-c will be compared between the standard of care arm and the inflammation-based treatment arm
% change in plasma HDL-c | 6 months
  Change in HDL-c will be compared between the standard of care arm and the inflammation-based treatment arm
% change in plasma triglycerides | 6 months
  Change in triglycerides will be compared between the standard of care arm and the inflammation-based treatment arm
% change in plasma high sensitivity C-reactive protein (hsCRP) | 6 months
  Change in hsCRP values will be compared between the standard of care arm and the inflammation-based treatment arm
% change in plasma IL-6 | 6 months
  Change in IL-6 values will be compared between the standard of care arm and the inflammation-based treatment arm
% change and absolute change in FAI-Score | 6 months
  Change in FAI-Score value will be compared between the standard of care arm and the inflammation-based treatment arm
% change and absolute change in CaRi-Heart Risk | 6 months
  Change in CaRi-Heart Risk value will be compared between the standard of care arm and the inflammation-based treatment arm
% change of FAI around identified individual coronary plaques | 6 months
  Change in FAI around identified individual coronary plaques will be compared between the standard of care arm and the inflammation-based treatment arm
FAI around identified individual coronary plaques | 6 months
  FAI around identified individual coronary plaques will be measured in both arms

CONTACTS AND LOCATIONS:
Overall Officials: Alexios S Antonopoulos, MD, PhD, Principal Investigator — 1st Cardiology Department, Hippokration General Hospital of Athens
Locations (1):
- 1st Cardiology Department, Hippokration General Hospital of Athens, Athens, Attica, Greece